CLINICAL TRIAL: NCT01231256
Title: A Study on Preventive Health Consultations in General Practice With Young Adults With Multiple Problems; a Randomised Controlled Study
Brief Title: Preventive Health Consultations With Young Adults With Multiple Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: North Denmark Region (Other Government); University of Aarhus (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Jørgen Lous, Professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: VN97/177
Record Dates: First submitted 2010-10-29; First posted 2010-11-01 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Quality of Life; Life Style
Keywords: Quality of life; preventive health consultation; General practice; resources; life style
MeSH Terms: interventions — Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- preventive health consultation (Experimental): Half participants randomized to a one hour preventive health consultation with their own general practitioner and a follow up consultation 3 months later
  Interventions: Behavioral: Preventive health consultation
- Control (No Intervention): Controls are not offered preventive health consultations, but had questionnaires as the intervention arm

INTERVENTIONS:
Behavioral: Preventive health consultation — A one hour preventive health consultation, based on completed baseline questionnaire, with one or two goal setting for a better life during the next year, with discussion and registration of resources, barriers, and time scheme. And a 3 month follow up consultation.
  Other Names: Consultation
  Arms: preventive health consultation

SUMMARY:
A new working method, i.e. a questionnaire completed at home followed by a patient-centred preventive health consultation with follow-up, can be used by all general practitioners (GPs) as a preventive offer to their patients with multiple problems in lifestyle, well-being or health behaviour, if this project is shown to be effective.

The investigators use a broad preventive offer in a structured way to young adults with multiple psychosocial problems (a certain risk profile) found by a screening questionnaire when arriving to the clinic.

The main hypothesis of the project is:

By using the questionnaire and subsequent patient-centred health consultation the GP is able to support the participants to improve their resources, their well-being and self-estimated health. Subsequently, relevant changes in health habits and life situation might be initiated in order to prevent or reduce future problems or illness.

DETAILED DESCRIPTION:
The main hypothesis of the project is:

By using the questionnaire and subsequent patient-centred health consultation the GP is able to contribute to improve the resources of the participants, their well-being and self-estimated health. Subsequently, relevant changes in health habits and life situation might be initiated in order to prevent or reduce future problems or illness.

The investigators want to test this hypothesis by describing

* the participating patients' situation at baseline (resources and problems), and after one year
* the content of the health interview (goals, resources and barriers for change)
* measure change of lifestyle and living conditions
* to evaluate the economic costs of the intervention
* evaluation of positive and negative effect of the health consultations for the patient and the GP

Partial hypothesis 1:

A large part of the target group experience many strains and have difficulties in fulfilling their personal expectations to a normal everyday life. Some might have risk behaviour.

The object of the project is to answer the following questions:

A. How is the baseline status of the participants (seven or more risk points) regarding self-estimated health, resources, family situation and risk score compared with the non-participants? (Paper 1)

B. Does the health consultation and follow-up consultation have effect within a year?

1. Initiate request for a change in behaviour within lifestyle and living conditions
2. Support a possible request for change by choosing one or two goals, as to somatic, mental and social issues
3. Contribute to an actual change in lifestyle and living conditions, in particular as regards to work, tobacco, alcohol, diet/weight and exercise
4. Contribute to a better self-estimated health
5. Contribute to improving resources.

Partial hypothesis 2:

The GP will in the project use a new working method that enables general impression and support of the individual's resources, which is very unlike the daily consultation, where the main focus is on risk thinking.

Does the registration by the GP and the patient reflect focus on improving resources?

1. Registration of resources and barriers to obtain the goals
2. Registration of time aspect to obtain these
3. Registration of need for further intervention (by GP or by others)

Partial hypothesis 3:

It has an effect to teach the GPs patient-centred preventive health consultation at short seminars/courses with focus on behavioural psychology, psychosocial medicine, and lifestyle issues such as tobacco, alcohol, drug abuse, diet / weight and exercise.

1. Have the GPs changed their view on preventive health consultations during the project period?
2. Have the GPs changed their view of changing potentials of their patients because of their participation in the study?

Method

Inclusion criteria for patients:

The practice secretary invites the patients to participate in the research project by asking all patients between 20-44 years coming to the clinic on a specific day or two in each month to complete a preliminary questionnaire (Screening questionnaire, SQ) asking 33 questions about lifestyle, resources, social situation and child problems. The quartile with most problems is invited to participate in the randomized trial. When five patients are included, no more patients are screened that day. The included patients receive a questionnaire (baseline questionnaire, BQ) of 23 pages they have to complete at home and return to the clinic as basis for the evaluation, the health consultation, and as a priming tool for the patient before the preventive health consultation.

Design The study is a randomized, controlled trial (RCT) with intervention (questionnaires and patient-centred preventive health consultations) compared with controls (questionnaires without health consultation). The intervention consisting of two consultations: the first of 60 minutes duration and follow-up of 20 minutes after three months. Both groups had postal follow-up questionnaires after one year.

Content of consultations is chosen by the patients, based on their completed questionnaires and own ideas of main problems, wishes and ability to improve their living conditions, health and quality of life guided and supported by the GP.

A follow-up after 3, 5 and 10 years is possible. Max 50 GPs can participate in the project with each max 20 health interviews (including a follow-up within three months) per year. That means approximately two interviews every month.

The inclusion period is expected to be about 1½ year from February 1998 to September 1999. A maximum of 1000 persons in the intervention group and 1000 in the control group can be included.

Randomisation When the BQ is returned to the clinic, the secretary makes a telephone block randomisation by phoning the project secretary, where every GP has a randomisation scheme with 40 computer-generated random numbers: 20 even numbers and 20 odd numbers to tick off in order when used. Patients hitting an even number will be offered a health interview, whereas patients with odd numbers will have to settle for the inspiration of the questionnaire and the regular visits to the GP. Both groups will be included in the follow-up schedule after a year, and possibly after 3, 5 and 10 years.

Inclusion criteria for GPs All 325 GPs in the county will be invited to a weekend course and offered the possibility to attend the project. If more than 50 GPs have registered for the project, the county is able to close for more registrations. The project team will organize and implement relevant courses. Firstly, all the county's GPs are invited to a course on 16 -17 January 1998 or 27-28/3-98 where senior school psychologist Per Kjeldsen, Aalborg, and clinical psychologist Annette Winter, Aarhus will teach and provide assignments based on different theories and behavioural problems. The project will be presented. Jens Tølbøll-Mortensen will teach about occupational medicine. Some meetings on factual knowledge about alcohol abuse, tobacco, the dietary importance, and cardiovascular diseases will be held. Furthermore, there will be follow-up courses during the project period about psychosocial preventive aspects on health and illness behaviour and the "health fraction".

Power calculation With a minimal relevant difference in Quality of life (SF12) of 3 (for example 47 and 50, and SD=10) and a type 1 error (alfa) of 0.05 and a type two error (1-beta) of 0.80, meaning that the investigators need 178 persons in each group.

Material A. The Screening questionnaire, SQ, consists of 33 problem questions within three main fields: family/social situation, resources and lifestyle. Most of the questions used are taken from different questionnaires used in other national and international studies, and some are constructed by KSF in accordance with psychosocial literature and 25 years experience as a GP. The number of problems is decisive for whether the patient will be included in the project or not. The quartile with most problems could be included. Some of the questions were binary and some had a five-graded answer category, where the three worst categories were defined as having a problem. After pilot-testing in four clinics the inclusion criteria were seven or more problems.

B. Baseline questionnaire, BQ consists of about 80 questions about family situation, resources, work, education, quality of life, health, disease and health behaviour, consumption of food, medicine, tobacco, alcohol and drugs. The BQ was based on the Danish population health and illness statistics every five years (Danish Institute of Clinical Epidemiology, DIKE), international studies, and a former study on preventive health consultations in Region North, Denmark. The 23-page questionnaire is to be completed by the patient at home.

C. In the last part of the health consultation the patient and the GP have to complete the dialogue chart (DC1), together, evaluating the health consultation's objectives, the patient's goals, and patient's resources, barriers and time needed to obtain these goals.

D. After the 3-month follow-up a similar DC2 was completed. E. A GP's evaluation form completed by the GP before and after the study. F. An intermediate telephone interview of the participating GPs by KSF. G. A one-year follow-up questionnaire, OQ is almost identical to the BQ questionnaire, but added a few final questions. The OQ questionnaire was mailed to both groups and completed at home, and returned to the project secretary by post.

Intervention elements

1. Courses for the GPs.
2. Questionnaires to the patients (interventions and controls). 2a. Screening questionnaire (SQ). 2b. Baseline questionnaire (BQ). 2c. One year questionnaire (OQ).
3. Health consultations with dialogue chart (DC1 and DC2).
4. Questionnaire and telephone interview with the GPs.

Financial support:

Department of Quality development, County of North Jutland, Lundbeck foundation, Fond for financing research in general practice and the health system in Denmark, PLU-foundation, Health Insurance Foundation, Sara Krabbes Legacy, University of Aarhus, University of Southern Denmark, University of Copenhagen,

ELIGIBILITY:
Inclusion Criteria:

* patients coming to the clinic
* having multiple problems (the quartile with most problems)

Exclusion Criteria:

* Do not want to participate
* Do not understand Danish well enough to complete the questionnaires
* Have too few problems
* Have severe psychiatric disease

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 495 (Actual)
Dates: Start 1998-02; Primary Completion 2001-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Quality of Life (SF12) | one year after intervention
  Change in Quality of Life one year after preventive health consultation (Physical Component (PCS) and Mental Component score (MCS))

SECONDARY OUTCOMES:
Change in life style | One year after intervention
  Smoking, diet, exercise, weight loss, acohol use
Change in self evaluated Health | one year after intervention
  Question about self evaluated health (on a five point scale)
Fraction with goal-setting | during the preventive health consultation
  Fraction with one or two goal-settings during the preventive health consultation
Change in problems with network | one year after preventive health consultation
  Problems with networking, four questions (from 0 to 4 problem-points each, total range 0 to 16 problem-points)
Change in resources | one year after preventive health consultation
  Problems with resources five questions (from 0 to 4 problem-points each, total range 0 to 20 problem-points)
Change in social problems | one year after preventive health consultation
  Social problems (i.e. unemployment, family problems, child problems, ect.). A total of 15 possible problems.
Written statements about own resources and barriers to obtain the chosen goal | during the preventive health consultation
  Quantitative and qualitative analysis of participants written statements about own resources and barrieres at the preventive health consultation and at follow up consultation after 3 months
Goals fulfilled after one year | one year after preventive health consultation
  Fraction of goals fulfilled after one year - analyses in relation to goal, resources and barriers, and status at baseline
Cost of the intervention | after one year
  Cost of the intervention seen in relation to outcomes
Side effects | after one year
  Registration of any side effects or harm during the study or in the questionnaires. Written statements by participants at one year follow-up, and by the GPs

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen Lous, Prof, DMSc, Study Director — University of Southern Denmark; Kirsten Freund, MD, GP, Principal Investigator — University of Southern Denmark
Locations (1):
- Research Unit for General Practice, University of Southern Denmark, Odense C, Denmark

REFERENCES:
- [Result] Freund KS, Lous J. [Potentially marginalized 20-44-years-olds in general practice. Who are they? The results of a questionnaire screening]. Ugeskr Laeger. 2002 Nov 11;164(46):5367-72. Danish. PMID 12469380
- [Result] Freund KS, Lous J. The effect of preventive consultations on young adults with psychosocial problems: a randomized trial. Health Educ Res. 2012 Oct;27(5):927-45. doi: 10.1093/her/cys048. Epub 2012 Apr 2. PMID 22473217
- [Result] Hansen E, Fonager K, Freund KS, Lous J. The impact of non-responders on health and lifestyle outcomes in an intervention study. BMC Res Notes. 2014 Sep 11;7:632. doi: 10.1186/1756-0500-7-632. PMID 25213806
- [Result] Lous J, Freund KS. Predictors of weight loss in young adults who are over-weight or obese and have psychosocial problems: a post hoc analysis. BMC Fam Pract. 2016 Apr 11;17:43. doi: 10.1186/s12875-016-0437-8. PMID 27068690